CLINICAL TRIAL: NCT01592032
Title: Concentration and Antibiotic Activity in Antibiotic Lock Solutions
Brief Title: Concentration of Antimicrobials in Catheter-lock Solutions
Acronym: CONAN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Navarrra Hospital (Clinica Universitaria) (Other)
Responsible Party: Principal Investigator, José Luis del Pozo, Medical Doctor, Ph. D., Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAS110775; 2010-023814-29 (EudraCT Number)
Record Dates: First submitted 2012-04-24; First posted 2012-05-04 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Catheter-Related Infections; Bacteremia.
Keywords: Antibiotic-lock technique.; In vivo antimicrobial concentration.; Antimicrobial bioactivity.
MeSH Terms: conditions — Catheter-Related Infections; Bacteremia | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vancomycin antimicrobial-lock (Experimental): Vancomycin antimicrobial-lock solution. Dosage: 2 mg/mL. Dosage form: liquid in syringe. Frequency: 1. Duration: from 1 to 10 days according to HPLC corrected by urea gradient.
  Interventions: Drug: Vancomycin antimicrobial-lock solution
- Teicoplanin antimicrobial-lock (Experimental): Teicoplanin antimicrobial-lock solution. Dosage: 10 mg/mL. Dosage form: liquid in syringe. Frequency: 1. Duration: from 1 to 10 days according to HPLC corrected by urea gradient.
  Interventions: Drug: Teicoplanin antimicrobial-lock solution
- Linezolid antimicrobial-lock (Experimental): Linezolid antimicrobial-lock solution. Dosage: 1.8 mg/mL. Dosage form: liquid in syringe. Frequency: 1. Duration: from 1 to 10 days according to HPLC corrected by urea gradient.
  Interventions: Drug: Linezolid antimicrobial-lock solution
- Daptomycin antimicrobial-lock (Experimental): Daptomycin antimicrobial-lock solution. Dosage: 5 mg/mL. Dosage form: liquid in syringe. Frequency: 1. Duration: from 1 to 10 days according to HPLC corrected by urea gradient.
  Interventions: Drug: Daptomycin antimicrobial-lock solution
- Tigecycline antimicrobial-lock (Experimental): Tigecycline antimicrobial-lock solution. Dosage: 4.5 mg/mL. Dosage form: liquid in syringe. Frequency: 1. Duration: from 1 to 10 days according to HPLC corrected by urea gradient.
  Interventions: Drug: Tigecycline antimicrobial-lock solution

INTERVENTIONS:
Drug: Vancomycin antimicrobial-lock solution — Randomization of 5 patients into vancomycin antimicrobial-lock solution arm for 1, 3, 5, 7 and 10 days according to HPLC corrected by urea gradient. The arm can be stopped any time from day 1 to day 10 in case of antimicrobial concentration less than 1 mg/mL.
  Other Names: vancomycin: vancomicina sala 500 mg vial.; sodium heparin 1%, 5000 IU/5ml.; sodium chloride 0,9% 10 ml vial.
  Arms: Vancomycin antimicrobial-lock
Drug: Teicoplanin antimicrobial-lock solution — Randomization of 5 patients into teicoplanin antimicrobial-lock solution arm for 1, 3, 5, 7 and 10 days according to HPLC corrected by urea gradient. The arm can be stopped any time from day 1 to day 10 in case of antimicrobial concentration less than 1 mg/mL.
  Other Names: teicoplanin: targocid 200 mg vial.; sodium heparin 1%, 5000 IU/5ml.; sodium chloride 0,9% 10 ml vial.
  Arms: Teicoplanin antimicrobial-lock
Drug: Linezolid antimicrobial-lock solution — Randomization of 5 patients into linezolid antimicrobial-lock solution arm for 1, 3, 5, 7 and 10 days according to HPLC corrected by urea gradient. The arm can be stopped any time from day 1 to day 10 in case of antimicrobial concentration less than 1 mg/mL.
  Other Names: linezolid: zyloxid 2 mg/ml, 300 ml vial.; sodium heparin 1%, 5000 IU/5ml.; sodium chloride 0,9% 10 ml vial.
  Arms: Linezolid antimicrobial-lock
Drug: Daptomycin antimicrobial-lock solution — Randomization of 5 patients into daptomycin antimicrobial-lock solution arm for 1, 3, 5, 7 and 10 days according to HPLC corrected by urea gradient. The arm can be stopped any time from day 1 to day 10 in case of antimicrobial concentration less than 1 mg/mL.
  Other Names: daptomycin: cubicin 350 mg vial.; sodium heparin 1%, 5000 IU/5ml.; lactated ringer´s solution 500 ml viaflo.
  Arms: Daptomycin antimicrobial-lock
Drug: Tigecycline antimicrobial-lock solution — Randomization of 5 patients into tigecycline antimicrobial-lock solution arm for 1, 3, 5, 7 and 10 days according to HPLC corrected by urea gradient. The arm can be stopped any time from day 1 to day 10 in case of antimicrobial concentration less than 1 mg/mL.
  Other Names: tigecycline: tygacil 50 mg vial.; sodium chloride 0,9% 10 ml vial.; sodium heparin 1%, 5000 IU/5ml.
  Arms: Tigecycline antimicrobial-lock

SUMMARY:
The antibiotic lock technique (ALT) is used as local treatment for Catheter-Related Bacteremia (CRB). It consists in the administration of a concentrated antimicrobial solution with a calculated volume to fill the lumen of the catheter. The lock solution is indwelled within the catheter for a defined period of hours or days before been removed.

Currently, the Infectious Diseases Society of America (IDSA) Guidelines for treatment and management of CRB, recommends to change the antibiotic solution every 24 hours.

The investigators expect to determine the stability of the concentration of vancomycin, teicoplanin, linezolid, daptomycin and tigecycline used in lock solutions, and thus to assay the optimal timeframe that the concentration of antibiotic used in lock solution keeps its in vivo antimicrobial activity.

Study Hypothesis: An antibiotic lock solution maintains in vivo concentration and antimicrobial activity for at least 10 days after its infusion inside a subcutaneous port catheter.

DETAILED DESCRIPTION:
Primary Objective: Assess the antimicrobial concentration of catheter-lock solutions at the end of port indwelling time. Secondary Objectives: 1) Assess bioactivity of antimicrobials in lock solutions at the end of port indwelling time. 2) Assess anticoagulant activity of antimicrobial-lock solutions at the end of port indwelling time.

Methods: Randomized, open, block allocation according to time of indwelling of the antimicrobial-lock within the ports, unicentric, clinical trial in patients older than 18 years old with a venous port implanted at Clínica Universidad de Navarra. Intevention: Randomization of 5 patients into one of five antimicrobial-lock solution arms for 1, 3, 5, 7 and 10 days according to HPLC corrected by urea gradient. Any study arm can be stopped at any time from day 1 to day 10, in case of antimicrobial concentration would be less than 1 mg/mL.

At the end of each antimicrobial lock time frame of ports (1, 3, 5, 7 and 10 days), the antimicrobial concentration will be determined by high performance liquid chromatography (HPLC) and corrected by urea gradient. The cut-off for the median antimicrobial concentration is 1 mg/mL.

ELIGIBILITY:
Inclusion Criteria:

* Intravenous access port recently inserted (≤ 3 days of insertion).
* Intravenous access port inserted more than 3 days before informed consent form signing patient. In this case, a blood sample from the catheter will be drawn for blood culture before administration of the antibiotic lock solution.
* Informed Consent Form Signed.

Exclusion Criteria:

* Patients with confirmed or suspected local or systemic infection related to the catheter.
* Reported allergy or intolerance to the antibiotic employed for study lock solutions.
* Patients receiving oral, intravenous or intramuscular antibiotic treatment at the moment of inclusion in the clinical trial.
* Patients receiving oral, intravenous or subcutaneous anticoagulant treatment, in a higher dose than the one used for venous thrombosis prophylaxis at the moment of inclusion in the clinical trial.
* Patients younger than 18 years old.
* Pregnant women or women in nursing period.
* Personal incapacity to subscribe the informed consent to participate in the clinical trial.

Patient Replacement Criteria:

All patients and/or their legal representatives will be inform that they can leave the clinical trial in whenever they wish to do it, without prejudice to their medical attention.

Also, according to the criteria of the principal investigator, a patient could be separated from the clinical trial. The reasons to separate a patient from the study and replace him/her are:

* Severe adverse reaction that could threat the life of the patient.
* Resolution of the patient or from his/her legal representative to abandon the study.
* No attend to the extraction visit date.
* Development of clinical inconveniences that may indicate to abandon the study in behalf of the patient.
* While antibiotic lock solution is within the port, manipulation or use of the port for administration of any kind of medication or fluid.
* Impossibility to extract 4 ml of the antibiotic lock solution from the port.
* Impossibility to extract 5 ml of peripheral blood sample at the moment of extraction of the antibiotic lock solution.
* Use of any of the prohibited medications during the antibiotic lock solution is inside the port.
* Intentionally wish of the patient in abandoning the study before or after antibiotic lock solution has been administered, or while the antibiotic lock solution is inside the port.

All patients who abandon the study or would be separated from the study for the exposed reasons, will be replaced for new candidates who fulfil the inclusion criteria and have signed the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial concentration of catheter-lock solutions at the end of port indwelling time. | 1 to 10 days

SECONDARY OUTCOMES:
Bioactivity of antimicrobials in lock solutions at the end of port indwelling time. | 1 to 10 days
Anticoagulant activity of antimicrobial-lock solutions at the end of port indwelling time. | 1 to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: JOSE L DEL POZO, MD. Ph. D., Principal Investigator — Clinica Universidad de Navarra; CESAR E BUSTOS, MD., Study Chair — Clinica Universidad de Navarra; AITZIBER AGUINAGA, Pharm. D., Study Chair — Clinica Universidad de Navarra; JOSE R YUSTE, MD. Ph.D., Study Chair — Clinica Universidad de Navarra; JOSE R AZANZA, MD. Ph.D., Study Chair — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Result] Del Pozo JL, Rodil R, Aguinaga A, Yuste JR, Bustos C, Montero A, Espinosa G, Garcia-Fernandez N. Daptomycin lock therapy for grampositive long-term catheter-related bloodstream infections. Int J Clin Pract. 2012 Mar;66(3):305-8. doi: 10.1111/j.1742-1241.2011.02830.x. PMID 22340450
- [Result] Del Pozo JL, Garcia Cenoz M, Hernaez S, Martinez A, Serrera A, Aguinaga A, Alonso M, Leiva J. Effectiveness of teicoplanin versus vancomycin lock therapy in the treatment of port-related coagulase-negative staphylococci bacteraemia: a prospective case-series analysis. Int J Antimicrob Agents. 2009 Nov;34(5):482-5. doi: 10.1016/j.ijantimicag.2009.06.020. Epub 2009 Aug 26. PMID 19713086
- [Result] del Pozo JL. Role of antibiotic lock therapy for the treatment of catheter-related bloodstream infections. Int J Artif Organs. 2009 Sep;32(9):678-88. doi: 10.1177/039139880903200918. PMID 19882553
- [Result] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Result] del Pozo JL, Patel R. The challenge of treating biofilm-associated bacterial infections. Clin Pharmacol Ther. 2007 Aug;82(2):204-9. doi: 10.1038/sj.clpt.6100247. Epub 2007 May 30. PMID 17538551
- [Result] Sherertz RJ, Boger MS, Collins CA, Mason L, Raad II. Comparative in vitro efficacies of various catheter lock solutions. Antimicrob Agents Chemother. 2006 May;50(5):1865-8. doi: 10.1128/AAC.50.5.1865-1868.2006. PMID 16641463
- [Result] Fennell JP, O'Donohoe M, Cormican M, Lynch M. Linezolid lock prophylaxis of central venous catheter infection. J Med Microbiol. 2008 Apr;57(Pt 4):534-535. doi: 10.1099/jmm.0.47665-0. PMID 18349379
- [Result] LaPlante KL, Mermel LA. In vitro activity of daptomycin and vancomycin lock solutions on staphylococcal biofilms in a central venous catheter model. Nephrol Dial Transplant. 2007 Aug;22(8):2239-46. doi: 10.1093/ndt/gfm141. Epub 2007 Apr 1. PMID 17403700
- [Result] Del Pozo JL, Alonso M, Serrera A, Hernaez S, Aguinaga A, Leiva J. Effectiveness of the antibiotic lock therapy for the treatment of port-related enterococci, Gram-negative, or Gram-positive bacilli bloodstream infections. Diagn Microbiol Infect Dis. 2009 Feb;63(2):208-12. doi: 10.1016/j.diagmicrobio.2008.10.004. Epub 2008 Nov 21. PMID 19026506
- [Result] Raad I, Hanna H, Jiang Y, Dvorak T, Reitzel R, Chaiban G, Sherertz R, Hachem R. Comparative activities of daptomycin, linezolid, and tigecycline against catheter-related methicillin-resistant Staphylococcus bacteremic isolates embedded in biofilm. Antimicrob Agents Chemother. 2007 May;51(5):1656-60. doi: 10.1128/AAC.00350-06. Epub 2007 Mar 12. PMID 17353249
- [Result] Robinson JL, Tawfik G, Saxinger L, Stang L, Etches W, Lee B. Stability of heparin and physical compatibility of heparin/antibiotic solutions in concentrations appropriate for antibiotic lock therapy. J Antimicrob Chemother. 2005 Nov;56(5):951-3. doi: 10.1093/jac/dki311. Epub 2005 Sep 9. PMID 16155063
- [Result] Labthavikul P, Petersen PJ, Bradford PA. In vitro activity of tigecycline against Staphylococcus epidermidis growing in an adherent-cell biofilm model. Antimicrob Agents Chemother. 2003 Dec;47(12):3967-9. doi: 10.1128/AAC.47.12.3967-3969.2003. PMID 14638511